CLINICAL TRIAL: NCT01728779
Title: Single-Arm Phase II Study of Stereotactic Body Radiation Therapy Concurrent With Nelfinavir for Oligometastases
Brief Title: Stereotactic Body Radiation With Nelfinavir for Oligometastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J12137; NA_00069585 (Other: JHMIRB)
Record Dates: First submitted 2012-10-12; First posted 2012-11-20 (Estimated); Results first posted 2021-04-23 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Oligometastases
MeSH Terms: interventions — Nelfinavir; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nelfinavir w/Stereotactic Body Radiation Therapy (SBRT) (Experimental): Patients with metastatic lesions of the lung, liver, or bone will be candidates for treatment. Within three weeks of the initial treatment planning, a 15 Gy dose (per lesion site) of SBRT will be administered. Prior to SBRT, patients will initiate Nelfinavir oral therapy twice daily for 7 days. Once SBRT is completed, the patient will repeat the same Nelfinavir therapy for an additional 7 days for a total of 14 days of treatment.
  Interventions: Drug: Nelfinavir; Radiation: Stereotactic Body Radiation (SBRT)

INTERVENTIONS:
Drug: Nelfinavir — Commercially available nelfinavir (1250 mg) will be administered orally twice daily for 14 days.
  Other Names: Viracept
Radiation: Stereotactic Body Radiation (SBRT) — 15 Gy dose (per lesion site) of SBRT will be administered
  Other Names: Stereotactic Body Radiation; SBRT

SUMMARY:
Patients with metastatic lesions of the lung, liver, or bone will be candidates for treatment. Within three weeks of the initial treatment planning, a 15 Gy dose (per lesion site) of SBRT will be administered. Prior to SBRT, patients will initiate Nelfinavir oral therapy twice daily for 7 days. Once SBRT is completed, the patient will repeat the same Nelfinavir therapy for an additional 7 days for a total of 14 days of treatment.

DETAILED DESCRIPTION:
The use of radiation therapy to treat metastatic tumors is well established and promising data are emerging with the use of SBRT for metastatic disease. However, the use of a single large fraction concurrent with a radiosensitizer as is being proposed is not of proven benefit. This investigation aims to confirm the safety and efficacy for SBRT used concurrently with a radiosensitizer in the setting of oligometastatic disease. The dose selected has been chosen with the belief that it is safe and effective based on prior experience with SBRT of lung cancer, pancreatic cancer and brain radiosurgery. All patients will be treated with a single fraction (per lesion site), targeted to the lesion concurrently with the radiosensitizer Nelfinavir.

On the basis of this preclinical evidence, we propose a phase II study of Nelfinavir combined with SBRT in patients with oligometastatic disease. Because the standard dose of Nelfinavir for HIV patients is known to be safe and does inhibit the phosphorylation of Akt and decrease tumor hypoxia, we propose to study this in conjunction with a 15 Gy dose of SBRT. Experience with single-fraction pulmonary and pancreas SBRT provides a useful dose for this trial. With published data establishing the relative safety of large single-fraction SBRT to the lungs and pancreas, we have decided to proceed to determine the safety of 15 Gy SBRT concurrently with the radiosensitizer Nelfinavir. Once this is established, we propose to continue to enroll more patients to the study at this dose to determine the efficacy of this type of therapy.

The proposed study represents an informed estimate based on current knowledge of SBRT doses and those administered in currently approved image-guided protocols (brain, base of skull, cervico-thoracic spine, pancreas and liver). This study will refine the current understanding of single fraction radiation tolerance for normal tissues, thereby making it possible to treat future patients more safely and aggressively.

ELIGIBILITY:
Inclusion Criteria

* Patient's tumor(s) to be treated is(are) ≤ 5.0 cm or ≤250 cm3
* Patient must have metastasis at one or more of the following sites: bone, liver, lymph node and/or lung. No more than five lesions will be treated.
* Histological confirmation of malignancy (primary or metastatic tumor).
* Patient may have any prior therapy allowed aside from having had prior radiotherapy to the treatment site (see exclusion criteria 5.2.3).
* Patient must be ≥ 18 years of age.
* Patient must have a life expectancy ≥ 9 months.
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Patient must have normal organ and marrow function.
* Patient must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study
* Patients receiving any other investigational agents
* Patient who has had any prior radiotherapy to the treatment site(s)
* Patients taking drugs that are contraindicated with nelfinavir, including any of the following:

Amiodarone, Quinidine, Rifampin, Dihydroergotamine, Ergonovine, Ergotamine, Methylergonovine, Hypericum perforatum (St. John's wort), Lovastatin, Simvastatin, Pimozide, Midazolam, Triazolam

* Women of child bearing potential who refuse to take a pregnancy test prior to treatment
* Participation in another concurrent treatment protocol while being treated on this protocol and through to 3 months after treatment on this protocol has ended
* Pregnant women
* Inability to understand the informed consent document
* Inability to sign the informed consent document
* Poor liver function suggestive of cirrhosis or steatohepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-01-08 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phuoc Tran, M.D., Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 38 patients were accrued between January 2014 and December 2015 with one who withdrew consent and 37 were included in the analysis.
Period: Overall Study
Arm/Group | Nelfinavir w/Stereotactic Body Radiation Therapy (SBRT)
Started | 38
Completed | 37
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 38 patients were enrolled but one patient withdrew consent. The analysis included a total of 37 patients.
Arm/Group | Nelfinavir w/Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 37
Age, Customized [Median (Full Range); unit: years] | 65 [35 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Freedom From Local Progression (FFLP)
Description: To determine the 6-month Freedom From Local Progression rate (measured as a percentage of participants) in participants treated with radiosensitizer nelfinavir used concurrently with 15 Gy of stereotactic body radiation therapy (SBRT) delivered in 1 fraction in patients with oligometastatic disease. FFLP is defined as the percent of participants who were free from progression at the 6 month time point.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nelfinavir w/Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 37
percentage of participants | 78.4 [61.4 to 88.5]

2. Secondary Outcome: Total Number of Adverse Events Experienced by Participants
Description: To assess the toxicity of the radiosensitizer Nelfinavir used concurrently with 15 Gy of stereotactic body radiation therapy (SBRT) delivered in 1 fraction (per lesion site) in patients with oligometastatic disease. Toxicity is assessed by the total number of adverse events based on Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: 1 year
Measure: Number; unit: adverse events
Arm/Group | Nelfinavir w/Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 37
adverse events
  Anorexia | 20
  Anxiety | 17
  Cough | 25
  Agitation | 3
  Alanine Amino Trans increased | 3
  Alkaline Phosphatase increased | 4
  Alopecia | 8
  ALT Increase | 3
  Anemia | 23
  Apnea | 3
  Aspartate Amino Trans increased | 2
  Ataxia | 1
  Bilirubin Increased | 3
  Bloating | 6
  Bronchial Infection | 1
  Bruising | 7
  Chills | 6
  Colonic obstruction | 1
  Concentration Impairment | 7
  Conjunctivitis | 2
  Constipation | 18
  Creatinine increased | 1
  Cytokine Release Syndrome | 1
  Dehydration | 4
  Depression | 15
  Dermatitis | 1
  Diarrhea | 31
  Dizziness | 11
  Dry Mouth | 14
  Dyspepsia | 13
  Dyspnea | 25
  Edema | 21
  Esophageal pain | 3
  Esophagitis | 5
  Fatigue | 32
  Fecal Incontinence | 4
  Fever | 1
  Gastritis | 3
  Headache | 12
  Hearing Loss | 1
  Hematuria | 3
  Hemaglobin Increased | 3
  Hemorrhoids | 12
  Hiccups | 2
  Hot Flashes | 4
  Hyperglycemia | 32
  Hyperkalemia | 4
  Hypernatremia | 1
  Hypertension | 1
  Hypoglycemia | 2
  Hypokalemia | 2
  Hyponatremia | 1
  Hypoxia | 1
  Insomnia | 1
  Lymphocyte absolute decreased | 22
  Malaise | 2
  Nausea | 23
  Neuralgia | 12
  White blood cells decreased | 22
  Weight Loss | 10
  Weight Gain | 15
  Vomitting | 10
  Urticaria | 2
  Urinary Incontinence | 25
  Urinary Frequency | 2
  Tremor | 3
  Toothache | 2
  Stomatitis | 2
  Stomach Pain | 11
  Oral mucositis | 3
  Perineal Pain | 1
  Periodontal Disease | 1
  Platelet count decreased | 13
  Proctitis | 2
  Pruritis | 9
  Radiation Recall Rctn | 3
  Rash | 2
  Skin Infection | 1
  Short term memory impairment | 1

3. Secondary Outcome: Percent of Lesions With Local Control at 6 Months Post-treatment
Description: To determine percent of lesions with local control at 6-months after SBRT delivered to a dose of 15 Gy in 1 fraction (per lesion site) combined with nelfinavir in patients with oligometastatic disease.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Nelfinavir w/Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 37
Number analyzed (Lesions) | 68
percentage of lesions | 76.5 [64.5 to 84.9]

4. Secondary Outcome: Participants' Clinical Progress While in Follow-up in Terms of Survival
Description: To assess the long-term clinical outcomes of this patient population after completion of SBRT in combination with Nelfinavir by determining the percentage of participants with Overall Survival (OS), Freedom From Distant Metastasis (FFDM) and the Progression-Free Survival (PFS).
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nelfinavir w/Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 37
percentage of participants
  Overall Survival | 90.7 [73.8 to 96.9]
  Freedom From Distant Metastasis | 62.4 [43.9 to 76.3]
  Progression-Free Survival | 57.6 [39.7 to 72]

5. Secondary Outcome: Quality of Life After Completion of Treatment
Description: To assess quality of life following completion of SBRT in combination with nelfinavir
Time Frame: 3 years
Population: Data was not collected for this outcome measure.
Arm/Group | Nelfinavir w/Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 0

6. Secondary Outcome: Phospho/ Akt Levels With Respect to Lesion Response
Description: Assess phospho-Akt protein in study participants to determine whether there is a correlation between the level protein and improved lesion response rate.
Time Frame: 3 months
Population: Data was not collected for this outcome measure.
Arm/Group | Nelfinavir w/Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 36 months.
Description: All AEs were recorded throughout the study, however there were only 5 grade 3 adverse events in three patients as defined by CTCAE.
Arm/Group | Nelfinavir w/Stereotactic Body Radiation Therapy (SBRT)
All-Cause Mortality (participants affected / at risk) | 3/37
Serious Adverse Events (participants affected / at risk) | 3/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nelfinavir w/Stereotactic Body Radiation Therapy (SBRT) (N=37)
Anxiety (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Weight Loss (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nelfinavir w/Stereotactic Body Radiation Therapy (SBRT) (N=37)
Anorexia (Psychiatric disorders) | 19 (19)
Anxiety (Psychiatric disorders) | 16 (16)
cough (Respiratory, thoracic and mediastinal disorders) | 24 (24)
Alopecia (General disorders) | 8 (8)
Anemia (Blood and lymphatic system disorders) | 22 (22)
Bilirubin (Renal and urinary disorders) | 9 (9)
Bloating (Gastrointestinal disorders) | 6 (6)
Bruising (General disorders) | 7 (7)
Chills (General disorders) | 6 (6)
Concentration impairment (Nervous system disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 18 (18)
Depression (Psychiatric disorders) | 15 (15)
Diarrhea (Gastrointestinal disorders) | 36 (36)
Dehydration (General disorders) | 4 (4)
Dizziness (Nervous system disorders) | 11 (11)
Dry mouth (General disorders) | 14 (14)
Dyspepsia (Gastrointestinal disorders) | 13 (13)
Dyspenea (General disorders) | 25 (25)
Edema (General disorders) | 21 (21)
Esophogitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Fatigue (General disorders) | 37 (37)
Fecal Incontinence (Gastrointestinal disorders) | 4 (4)
Headache (Nervous system disorders) | 12 (12)
Hemmorhoids (Gastrointestinal disorders) | 12 (12)
Hot Flashes (Endocrine disorders) | 4 (4)
Hyperglycemia (Endocrine disorders) | 32 (32)
Hyperkalemia (Blood and lymphatic system disorders) | 4 (4)
Lymphocyte Absolute Increase (Blood and lymphatic system disorders) | 37 (37)
Nausea (Gastrointestinal disorders) | 22 (22)
Neuralgia (Nervous system disorders) | 12 (12)
WBC Decrease (Blood and lymphatic system disorders) | 22 (22)
Vomitting (Gastrointestinal disorders) | 10 (10)
Weight Loss (General disorders) | 9 (9)
Weight Increase (General disorders) | 15 (15)
Urinary Incontinence (Renal and urinary disorders) | 25 (25)
Stomach Pain (General disorders) | 11 (11)
Platelet Count Decrease (Blood and lymphatic system disorders) | 13 (13)
Pruritis (General disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT01728779/Prot_SAP_000.pdf